CLINICAL TRIAL: NCT00440895
Title: A Randomized Trial of Early Discharge After Trans-Radial Stenting of Coronary Arteries in Acute Myocardial Infarction and RESCUE-PCI: The EASY-RESCUE Pilot Study
Brief Title: A Randomized Trial of Early Discharge After Trans-radial Stenting of Coronary Arteries in Acute MI and Rescue-PCI
Acronym: EASY-RESCUE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Olivier F. Bertrand (Other)
Collaborators: Eli Lilly and Company (Industry); Cordis US Corp. (Industry)
Responsible Party: Sponsor-Investigator, Olivier F. Bertrand, MD PhD, Laval University
Organization: Laval University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EASY-RESCUE
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Myocardial Infarction; Ischemia
Keywords: Coronary artery stenting; Trans-radial; Intracoronary; Rescue-PCI
MeSH Terms: conditions — Myocardial Infarction; Ischemia | interventions — Abciximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 intracoronary + infusion (Experimental): Bolus abciximab i.c. (0.25 mg/kg) followed by 12 h infusion at 0.125 µg/kg/min (max 10µg/min).
  Interventions: Drug: Abciximab
- 2 intravenous (Active Comparator): Bolus abciximab i.v. (0.25 mg/kg) followed by 12 h infusion at 0.125 µg/kg/min (max 10µg/min).
  Interventions: Drug: Abciximab
- 3 Placebo (Placebo Comparator): Bolus of placebo followed by 12 h infusion (placebo).
  Interventions: Drug: Abciximab

INTERVENTIONS:
Drug: Abciximab — Abciximab (bolus) i.c. or i.v. or placebo, bolus dose is calculated according to current dosage (0.25 mg/kg) followed by 12 h infusion at 0.125 µg/kg/min (max 10µg/min).
  Other Names: Abciximab (ReoPro)

SUMMARY:
* Abciximab administration is safe and reduces ischemic complications in patients undergoing rescue PCI after failed thrombolysis compared to placebo.
* Abciximab improves angiographic scores and ventricular function after rescue-PCI compared to placebo.
* Intracoronary abciximab administration is more effective than intravenous route of administration in terms of acute and mid-term angiographic and clinical results.
* Intracoronary and intravenous bolus administration of abciximab dose provides similar platelet aggregation inhibition (PAI).
* There is a significant relationship between PAI after abciximab administration and indexes of myocardial perfusion.
* Routine use of Sirolimus-eluting stents (Cypher, Cordis, US) in rescue-PCI is associated with a low rate of target vessel revascularization.
* Cardiac MRI early and late after rescue-PCI provides detailed information on myocardial injury and irreversible necrosis, which are correlated with angiographic perfusion scores.
* After uncomplicated trans-radial rescue PCI, patients can be retransferred early to their referring center.

DETAILED DESCRIPTION:
OBJECTIVES AND END-POINTS

The objectives of the present pilot study are to assess 1) the benefits and safety of abciximab i.c. or i.v. compared to placebo in rescue PCI and trans-radial approach, 2) the relationship between platelet aggregation inhibition and perfusion scores and to demonstrate 3) better perfusion scores with i.c. abciximab as compared to i.v. abciximab or placebo.

The Primary ANGIOGRAPHIC end-point will be the TIMI score and myocardial blush grade after rescue-PCI at baseline and at 6-months follow-up.

The Secondary CLINICAL end-point will be:

* the composite of death, stroke, repeat-myocardial infarction, urgent target vessel revascularization and major bleedings at 30 days after rescue PCI.
* composite of death, repeat-myocardial infarction, repeat target vessel revascularization at 6 months following rescue PCI.

The Secondary PLATELETS end-point will be the proportion of patients with platelet aggregation inhibition ≥ 95% and mean platelet aggregation inhibition 10 minutes post-bolus administration.

The Secondary ANGIOGRAPHIC end-points will be the angiographic late loss and the restenosis rate (Diameter stenosis ≥ 50%) in the culprit artery.

Other exploratory end-points include the feasibility and safety of early transfer to the referring hospital after uncomplicated primary PCI, cardiac MRI measurements and PAI 6 hr after bolus administration.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acute myocardial infarction eligible for rescue PCI within 24 hrs of symptoms.
* Failed thrombolysis (defined as less than 50% reduction of ST-elevation at 90 min ECG in the lead with previous maximal ST-segment elevation).
* Patient > 18 years old.
* Patient and treating interventional cardiologist agree for randomization.
* Patient will be informed of the randomization process and will sign an informed consent.
* Diagnostic and therapeutic intervention performed through transradial/transulnar approach.
* The culprit lesion in a native coronary artery can identified and is suitable for immediate angioplasty and stent implantation.

Exclusion Criteria:

* Age > 75 years old
* Body weight < 65 kg
* Concurrent participation in other investigational study
* Intolerance or allergy to ASA, clopidogrel or ticlopidine precluding treatment for 12 months
* Any significant blood dyscrasia, diathesis or INR > 2.0.
* Any clinical contraindication to abciximab administration i.e. known structural intracranial lesion, thrombocytopenia (< 100,000), hemoglobin level < 10 g/dl
* Patient has received more than one dose of thrombolytic within 24 hours of symptoms
* Previous treatment with glycoproteins IIb-IIIa inhibitors within 30 days
* Perceived increased risk of intracranial or severe bleeding i.e. previous stroke/TIA, alteration of consciousness, recent trauma or major surgery.
* Uncontrolled high blood pressure i.e. systolic blood pressure ≥ 180 mmHg and/or diastolic blood pressure ≥ 100 mmHg.
* Life expectancy less than 6 months owing to non-cardiac cause
* Evident cardiogenic shock

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-02; Primary Completion 2012-10 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
TIMI score and myocardial blush grade after rescue-PCI at baseline and at 6-month follow-up | 6 months

SECONDARY OUTCOMES:
1 Composite of death, stroke, repeat-MI, urgent target vessel revascularization and major bleedings at 30 days after rescue PCI | 1 month
2 Composite of death, repeat-MI, repeat target vessel revascularization at 6 months following rescue PCI | 6 months
3 Proportion of patients with platelet aggregation inhibition ≥ 95% and mean platelet aggregation inhibition 10 min post-bolus administration | 10 min post PCI
4 Angiographic late loss and restenosis rate (diameter stenosis ≥ 50%) in the culprit artery | 6 months
5 Exploratory end-points include the feasibility and safety of early transfer to the referring hospital after uncomplicated primary PCI, cardiac MRI measurements and PAI 6 h after bolus administration | 6-hr post PCI to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Olivier F Bertrand, MD, PhD, Principal Investigator — Laval Hospital Research Center
Locations (1):
- Laval Hospital, Québec, Quebec, Canada